CLINICAL TRIAL: NCT03471182
Title: Investigation of Cocaine Addiction Using mGluR5 PET and fMRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patrick Worhunsky, Assistant Professor of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000021196; 1K01DA042998-01A1 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-03-20 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence; Cocaine Addiction
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Psychiatry; Neuropsychological Tests; Cocaine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Psychiatric and Cognitive Testing (Active Comparator): All participants will complete psychiatric assessment and cognitive testing.
  Interventions: Behavioral: Psychiatric and Cognitive Testing
- Cocaine Self-adminstration (Active Comparator): This arm plans to assess the subjective (e.g., euphoric) and behavioral effects (e.g., self-administration) of cocaine in experienced, non-treatment seeking users of the drug in a human laboratory study of self-regulated cocaine administration.
  Interventions: Drug: Cocaine Self-adminstration
- Positron Emission Tomography (Active Comparator): All participants will complete a PET scan to assess mGluR5 receptors using [18-F]FPEB
  Interventions: Radiation: Positron Emission Tomography
- Magnetic Resonance Imaging (Active Comparator): All participants will complete one MRI scan to assess brain structure and function.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Behavioral: Psychiatric and Cognitive Testing — Interviews, questionnaires, and computer testing.
  Arms: Psychiatric and Cognitive Testing
Drug: Cocaine Self-adminstration — The intervention will include a training and safety session that consists of physician/nurse-administered cocaine followed by a self-regulated cocaine administration period under carefully controlled and closely monitored conditions.
  Other Names: cocaine hydrochloride
  Arms: Cocaine Self-adminstration
Radiation: Positron Emission Tomography — PET scans will be performed on a High Resolution Research Tomograph (HRRT), the highest resolution human brain scanner available. Antecubital venous catheters will be used for IV administration of the radiotracer and for venous blood sampling. A radial artery catheter may also be inserted by an experienced physician before the PET scan. At the beginning of each scan, the participants's head will be immobilized and a 6-minute transmission scan, using an orbiting 137Cs point-source, is obtained and used for attenuation correction. PET scans will be acquired using bolus or bolus plus constant infusion administration of [18F]FPEB.
  Other Names: PET
  Arms: Positron Emission Tomography
Other: Magnetic Resonance Imaging — Structural and functional MRI data will be acquired using a Siemens Trio TIM 3.0T system at the Yale Magnetic Resonance Research Center. High-resolution structural MRI data will be acquired to facilitate analysis of PET data and may be used in additional analysis of tissue volume and brain structure. Resting-state and task-based functional MRI data will be acquired using state-of-the-art multiband echo-planar imaging (EPI) gradient-echo sequences. Diffusion-weighted MRI data will also be acquired using multiband imaging sequences to investigate anatomical connectivity.
  Other Names: MRI, functional MRI
  Arms: Magnetic Resonance Imaging

SUMMARY:
The proposed research program will investigate the changes in brain chemistry and circuitry that 're-wire' the brain during chronic cocaine use, promote relapse, and complicate treatment efforts. Currently-using and non-treatment-seeking individuals with a cocaine use disorder will undergo a cocaine self-administration paradigm 2-5 days prior to completing positron emission tomography (PET) and functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Cocaine use disorder (CUD) remains a significant public health concern that is resistant to current treatments. Challenges to treating CUD include an imbalance in neurobiological systems that 're-wire' the brain such that appetitive and habitual processes influence decision-making and behavior. This research project aims to provide insight into this reorganized circuitry in CUD by investigating neurofunctional systems related to glutamatergic plasticity and functional brain networks during initial (2-5 days) abstinence. To target this potentially critical period of recovery, currently-using and non-treatment-seeking individuals with CUD will undergo a cocaine self-administration paradigm 2-5 days prior to completing [18F]FPEB positron emission tomography (PET) and functional magnetic resonance imaging (fMRI). Healthy comparison (HC) subjects that have participated in [18F]FPEB PET as part of other Yale approved protocols will be recruited to participate in the fMRI portion of this study.

Aim 1: To determine the availability of mGluR5 using [18F]FPEB PET during initial abstinence in individuals with CUD. The investigators hypothesize individuals with CUD, relative to HC, will exhibit concurrently and regionally specific increases (e.g., in the striatum) and decreases (e.g., in the prefrontal cortex) in mGluR5 availability.

Aim 2: To determine patterns of resting-state, response-inhibition, an automaticity related connectivity within and between large-scale functional networks using fMRI during initial abstinence in individuals with CUD. The investigators hypothesize network-based analyses of fMRI will reveal lower frontoparietal and greater limbic network modulation in CUD as compared to HC.

Aim 3: To explore the relationships between mGluR5 availability and functional network activity during initial abstinence in individuals with CUD. The investigators will perform multi-modal analysis of PET and fMRI data to examine links between molecular and functional systems in CUD using emerging 'fusion' approaches. While exploratory in nature, the investigators expect to find links between alterations in mGluR5 systems and functional reorganization in CUD (e.g., greater dorsostriatal mGluR5 may be linked to blunted frontoparietal inhibition).

Aim 4: To explore the relationships between mGluR5 availability, functional network activity (and their linkages) with cocaine self-administration, disease severity and chronicity, and psychometric assessments of impulsivity and compulsivity. While exploratory in nature, the investigators expect more substantial neurofunctional alterations during initial abstinence will be associated with greater cocaine self-administration, disease severity, impulsivity and compulsivity in individuals with CUD.

ELIGIBILITY:
Inclusion Criteria:

* All participants:

  * Age 21 - 60 years
  * Provide voluntary, written, informed consent
  * Physically healthy by medical history, physical, neurological, ECG, and laboratory examinations
  * For females: non-lactating, no longer of child-bearing potential or agreeing to practice effective contraception during the study (e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine system [IUS]; barrier methods: condom or occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository; male partner sterilization; true abstinence when this is in line with the preferred and usual lifestyle of the subject), and a negative serum pregnancy test
* Participants with a cocaine use disorder:

  * DSM-5 criteria for moderate or severe cocaine-use disorder
  * Recent street cocaine use in excess of quantities used in the current study
  * Intravenous and/or smoked (crack/freebase) cocaine use
  * Positive urine toxicology screen for cocaine
* Healthy comparison participants:

  * Successful completion of an [18F]FPEB scan as part of another Yale approved protocol as a healthy control/comparison subject

Exclusion Criteria:

* All participants:

  * Any condition that, in the opinion of investigators, would prevent compliance with the study protocol
  * A history of significant medical or neurological illness (e.g., coronary artery disease, significant anemia, seizures)
  * Current use of psychotropic and/or potentially psychoactive medications
  * Physical or laboratory evidence of pregnancy
  * Meet any additional PET/MR imaging-related exclusion criteria, including:
  * Presence of MRI incompatible implants and other contraindications for MRI (e.g., pacemaker, artificial joints, non-removable body piercings, etc.)
  * Participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the participant to exceed the yearly dose limits
  * History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).
  * Claustrophobia
  * Severe motor problems that prevent the subject from lying still for PET/MR imaging
  * Complaints of chronic pain (e.g., as the result of rheumatoid arthritis)
  * Current, past or anticipated exposure to radiation in the work place
* Participants with a cocaine use disorder:

  * Other drug use disorder (except for tobacco-use disorder)
  * Less than 1 year of cocaine use disorder
  * A DSM-5 major psychiatric diagnosis (schizophrenia, bipolar disorder, etc.) unrelated to cocaine
* Healthy comparison participants:

  * Any DSM-5 major psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), except tobacco-use disorder
  * Positive drug screen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Worhunsky, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with NIH Grants Policy on Sharing of Unique Research Resources, including the "Sharing of Biomedical Research Resources: Principles and Guidelines for Recipients of NIH Grants and Contracts" (December, 1999), all research resources generated will be freely distributed, as available, to appropriate, qualified academic investigators for non-commercial research purposes. All data will be de-identified before sharing, using procedures in compliance with HIPPA and Yale Human Investigation Committee standards. No available data sets or supporting information will contain subject names, addresses or other specific personal identification.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: In accordance with institutional standards and guidelines, after termination of this study and completion of all analysis and publications, all data and screening information will be anonymized and kept in a secure fashion for the purpose of further analyses indefinitely unless prevailing University or Federal guidelines at the time require a change.
Access Criteria: In accordance with institutional standards and guidelines, researchers must submit a requisition form that describes their specific hypotheses and details specific data or supporting information being requested. Requests will be reviewed by senior study personnel.

REFERENCES:
- [Derived] Kohler RJ, Zhornitsky S, Potenza MN, Yip SW, Worhunsky P, Angarita GA. Cocaine self-administration behavior is associated with subcortical and cortical morphometry measures in individuals with cocaine use disorder. Am J Drug Alcohol Abuse. 2024 May 3;50(3):345-356. doi: 10.1080/00952990.2024.2318585. Epub 2024 Mar 29. PMID 38551365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the New Haven, CT community, through current/past enrollment in similar research at the Cocaine Research Clinic and Yale PET Center as well as through community advertising (e.g., flyers). The first participant was enrolled on February 26, 2018 and the last participant was enrolled on June 30, 2022.
Pre-assignment Details: Of 32 enrolled individuals, 17 met inclusion criteria for participants with cocaine-use disorder and 8 met criteria as healthy-comparison participants. Twenty historical healthy-comparison participants were not considered enrolled in this study.
Groups:
- Adults With a Cocaine-use Disorder (CUD): Non-treatment-seeking, medically healthy adults meeting DSM-5 criteria for a moderate or severe cocaine-use disorder.
- Healthy Comparison Adults, MRI (HC-MRI): Medically and psychologically healthy adults enrolled in this study to complete the magnetic resonance imaging (MRI) procedures as part of a comparison Group to examine MRI Outcome Measures.
- Historical Healthy Comparison Adults, PET (HHC-PET): A historical sample of medically and psychologically healthy adults completing positron emission tomography (PET) procedures. This sample was compiled uniquely for this study from a larger set of historical data to form a comparison Group to examine PET Outcome Measures.
Period: Overall Study
Arm/Group | Adults With a Cocaine-use Disorder (CUD) | Healthy Comparison Adults, MRI (HC-MRI) | Historical Healthy Comparison Adults, PET (HHC-PET)
Started | 17 | 8 | 20
Completed MRI Procedures | 16 | 7 | 0
Completed PET Procedures | 15 | 0 | 0
Completing Both MRI and PET | 14 | 0 | 0
Completed | 14 | 7 | 20
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Technical failure | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In addition to participants enrolled in this study (N=17 CUD, N=8 HC-MRI), baseline characteristics are provided for the sample of comparison adults completing PET procedures (N=20 HC-PET) as part of other studies.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults With a Cocaine-use Disorder (CUD) | Healthy Comparison Adults, MRI (HC-MRI) | Historical Healthy Comparison Adults, PET (HHC-PET) | Total
Number analyzed (Participants) | 17 | 8 | 20 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (6.5) | 36.6 (4.8) | 49.0 (7.4) | 46.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 7 | 13
  Male | 12 | 7 | 13 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 15 | 8 | 19 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 8 | 17
  White | 9 | 5 | 12 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 8 | 20 | 45
Positive toxicology screen indicating recent cocaine use [Count of Participants; unit: Participants] — Standard commercially available urinalysis cups were used to test for commonly used substances including cocaine, amphetamines, marijuana, opiates, benzodiazepines, and barbiturates. Tests were performed to confirm recent cocaine use in participants with a CUD and the absence of drug use in HC participants.
  Participants | 17 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Regional Availability of Metabotropic Glutamate Type-5 Receptors (mGluR5)
Description: Receptor availability assessed as the volume of distribution (VT) of [18F]FPEB radiotracer, measured using positron emission tomography (PET). Higher [18F]FPEB VT values indicate a greater availability of mGluR5 receptors.
Time Frame: Following 2-5 days of cocaine abstinence
Population: Standard analysis of PET data requires a high-resolution MRI image for anatomical localization; thus only participants with a CUD completing both PET and MRI procedures(N=14 CUD) were analyzed. PET data was not collected on the Group healthy comparison adults completing only MRI procedures (HC-MRI).
Measure: Mean (Standard Deviation); unit: mL*cm^3
Arm/Group | Adults With a Cocaine-use Disorder (CUD) | Historical Healthy Comparison Adults, PET (HHC-PET)
Number analyzed (Participants) | 14 | 20
mL*cm^3
  Ventral striatum | 36.48 (8.05) | 32.19 (5.58)
  Caudate | 25.67 (7.29) | 22.41 (4.75)
  Putamen | 30.31 (5.84) | 26.06 (5.26)
  Orbitofrontal cortex | 30.40 (6.13) | 26.36 (4.61)
  Anterior cingulate cortex | 32.54 (6.88) | 28.73 (5.54)
  Ventromedial prefrontal cortex | 33.95 (7.21) | 29.41 (5.34)
  Inferior frontal gyrus | 28.42 (6.08) | 24.78 (4.25)
  Middle frontal gyrus | 28.37 (6.94) | 24.95 (4.36)
  Superior frontal gyrus | 27.55 (6.33) | 23.65 (4.30)
Statistical Analysis 1: Comparison: Adults With a Cocaine-use Disorder (CUD) vs Historical Healthy Comparison Adults, PET (HHC-PET); Outcome Measure Data were tested using a single linear mixed effects model. The 9 regions of interest (i.e., all 9 Rows of the Outcome Measure Data) were included in the model as a within-subjects factor for the fixed-effect of region. Group (i.e., CUD, HHC-PET) was included in the model as a between-subjects factor for the fixed-effect of group. The model also included the region-by-group interaction term and a factor to model the random-effect of participant; Test type: Superiority; p = 0.035, Mixed Models Analysis — Primary hypothesis of a group difference (i.e., CUD vs HHC-PET participants) in mGluR5 availability was assessed as the significance level of the fixed-effect of group at a threshold of p<0.05

2. Primary Outcome: Functional Brain Network Engagement Associated With Response Inhibition
Description: Independent component analysis (ICA) of functional MRI data separates brain activity associated with distinct functional networks. Comparing the activity in these networks to the fMRI task events using a regression analysis produces a beta-weight where a larger beta indicates the network was more activated or 'engaged' in processing the task demands. In this study, participants completed a Go/NoGo task to assess brain processing associated with infrequent-stimulus response inhibition (i.e., correct NoGo's) compared to frequent-stimulus responses (i.e., correct Go's).
Time Frame: Following 2-5 days of cocaine abstinence.
Population: All participants who performed a Go/NoGo task during MRI procedures. Functional MRI data of Go/NoGo performance was not collected on the Group historical healthy comparison adults who had completed PET procedures (HHC-PET).
Measure: Mean (Standard Error); unit: Unitless beta coefficient
Groups:
- Healthy Comparison Adults, MRI (HC-MRI): Medically and psychologically healthy comparison adults completing magnetic resonance imaging (MRI) procedures as part of this study.
Arm/Group | Adults With a Cocaine-use Disorder (CUD) | Healthy Comparison Adults, MRI (HC-MRI)
Number analyzed (Participants) | 16 | 7
Unitless beta coefficient
  Right frontoparietal network | 0.409 (0.103) | 0.125 (0.156)
  Left frontoparietal network | 0.349 (0.159) | 0.037 (0.241)
  Basal ganglia network | 0.175 (0.103) | -0.240 (0.156)
  Cingulo-insula network | 0.103 (0.121) | -0.271 (0.183)
Statistical Analysis 1: Comparison: Adults With a Cocaine-use Disorder (CUD) vs Healthy Comparison Adults, MRI (HC-MRI); Test type: Superiority — Outcome Measure Data were tested using a single linear mixed effects model. The 4 brain networks of interest (i.e., all 4 Rows of the Outcome Measure Data) were included in the model as a within-subjects factor for the fixed-effect of network. Group (i.e., CUD, HC-MRI) was included in the model as a between-subjects factor for the fixed-effect of group. The model also included the network-by-group interaction term and a factor to model the random-effect of participant; p = 0.024, Mixed Models Analysis — Primary hypothesis of group differences (i.e., CUD vs HC-MRI participants) in functional brain network engagement was assessed as the significance level of the fixed-effect of group at a threshold of p<0.05

3. Primary Outcome: Resting-state Functional Brain Network Activity, Fractional Amplitude of Low-frequency Fluctuations (fALFF)
Description: Independent component analysis (ICA) of functional MRI data separates brain activity associated with distinct functional networks. The fractional amplitude of low-frequency fluctuations (fALFF) during resting-state reflects a measure of the general health status of a network, comprised of both the strength of network activity and within-network connectivity absent of any specific cognitive demands.
Time Frame: Following 2-5 days of cocaine abstinence.
Population: Participants who completed resting-state functional MRI procedures. Two the 16 CUD participants completing MRI were excluded from analysis due to insufficient data and poor image quality resulting from excessive head motion. Resting-state functional MRI data were not available on the Group historical healthy comparison adults who had completed PET procedures (HHC-PET).
Measure: Mean (Standard Error); unit: Unitless ratio
Arm/Group | Adults With a Cocaine-use Disorder (CUD) | Healthy Comparison Adults, MRI (HC-MRI)
Number analyzed (Participants) | 14 | 7
Unitless ratio
  Default-mode network | 0.747 (0.021) | 0.726 (0.030)
  Right frontoparietal network | 0.749 (0.019) | 0.772 (0.026)
  Left frontoparietal network | 0.739 (0.021) | 0.734 (0.030)
  Basal ganglia network | 0.636 (0.036) | 0.590 (0.051)
  Cingulo-insula network | 0.707 (0.029) | 0.726 (0.041)
Statistical Analysis 1: Comparison: Adults With a Cocaine-use Disorder (CUD) vs Healthy Comparison Adults, MRI (HC-MRI); Outcome Measure Data were tested using a single linear mixed effects model. The 5 brain networks of interest (i.e., all 5 Rows of the Outcome Measure Data) were included in the model as a within-subjects factor for the fixed-effect of network. Group (i.e., CUD, HC-MRI) was included in the model as a between-subjects factor for the fixed-effect of group. The model also included the network-by-group interaction term and a factor to model the random-effect of participant; Test type: Superiority; p = 0.870, Mixed Models Analysis — Primary hypothesis of group differences (i.e., CUD vs HC-MRI participants) in fALFF was assessed as the significance level of the fixed-effect of group at a threshold of p<0.05

ADVERSE EVENTS:
Time Frame: Less than 30 days, typically 1-2weeks
Description: The group of Historical Healthy Comparison adults completing PET procedures during participation in other studies (HHC-PET) were monitored for Adverse Events by their original studies.
Arm/Group | Adults With a Cocaine-use Disorder (CUD) | Healthy Comparison Adults, MRI (HC-MRI)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/8
Other Adverse Events (participants affected / at risk) | 0/17 | 0/8

LIMITATIONS AND CAVEATS:
This study was greatly impacted by a COVID-related suspension in research activities and subsequent restrictions on facility operations. This resulted in lower participation and study adjustments including the discontinuation of cocaine self-administration procedures, the use of historical HC-PET data, and the collection of an HC-MRI sample (no HC completed both PET and fMRI). These alterations limit the statistical power of primary outcomes and the ability to perform planned secondary analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT03471182/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT03471182/ICF_001.pdf